CLINICAL TRIAL: NCT01061502
Title: Efficacy of the PROCELLERA Wound Dressing in the Healing of Skin Graft Donor Sites
Brief Title: Efficacy Study of a Bioelectric Dressing to Treat Skin Graft Donor Site Wounds
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vomaris Innovations (Industry)
Responsible Party: Andrew Blount, MD, Spectrum Health Blodgett Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: XSMP-014
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Burns; Wound Healing
Keywords: Burns; Wounds and Injuries; Skin Grafts, Bioelectric; Grafting, skin
MeSH Terms: conditions — Burns; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Procellera Wound Dressing (Experimental): Dressing indicated for partial and full-thickness wounds. Dressing changes every 5-7 days, more frequently if needed
  Interventions: Device: Procellera (Bioelectric Wound Dressing)
- Opsite Transparent Adhesive Dressing (Active Comparator): Polyurethane film dressing. Dressing changes every 5-7 days, more frequently if needed
  Interventions: Device: Opsite (Transparent Adhesive Dressing)

INTERVENTIONS:
Device: Procellera (Bioelectric Wound Dressing) — Dressing used on one-half of the donor graft site. Dressing changes every 5-7 days, more frequently if needed
  Other Names: Procellera; PROSIT; Procellera Wound Dressing; Procellera Device
  Arms: Procellera Wound Dressing
Device: Opsite (Transparent Adhesive Dressing) — Semi-occlusive wound dressing placed on one-half of the skin graft donor site. Dressing change every 5-7 days, more frequently if needed.
  Other Names: Opsite Dressing
  Arms: Opsite Transparent Adhesive Dressing

SUMMARY:
The purpose of this study is to determine whether the use of a bioelectric wound dressing is effective in the healing of skin graft donor site wounds.

ELIGIBILITY:
Inclusion Criteria:

* Wounds resulting from skin graft
* Split thickness wound
* Wound size greater than 2x2 cm
* Wounds must be ≥5 cm away from all other wounds
* Participant agrees to participate in follow-up evaluation
* Participant must be able to read and understand informed consent, and sign the informed consent

Exclusion Criteria:

* Concurrent participation in another clinical trial that involves an investigational drug or device that would interfere with this study
* Participant is to receive another topical antimicrobial agent other than the study dressing
* Participant with sensitivity or adverse reactions to silver or zinc
* Pregnancy or nursing an infant or child
* Immunosuppression
* Active or systemic infection
* Peripheral vascular occlusive disease
* Collagen vascular disease
* Connective tissue disease
* Participant undergoing active cancer chemotherapy
* Chronic steroid use
* Decision impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To compare epithelialization over time | 3 months

SECONDARY OUTCOMES:
To compare patient reported perception of pain | 3 months
To compare scarring | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew L Blount, MD, Principal Investigator — Blodgett Hospital; Richard Wilcox, MD, Study Director — Blodgett Hospital
Locations (1):
- Blodgett Hospital, Grand Rapids, Michigan, United States